CLINICAL TRIAL: NCT04008407
Title: Endoscopic Submucosal Dissection for Sessile Polyps and Laterally Spreading Lesions of the Colorectum Using a Selective Strategy - a Prospective Cohort Study
Brief Title: ESD for Colorectal LSL Using a Selective Strategy - a Prospective Cohort Study
Acronym: COVERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Director of Endoscopy, Western Sydney Local Health District
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU RED HREC/17/WMEAD/497
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Neoplasm; Endoscopic Mucosal Resection
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Intervention Model Description: Selective treatment algorithm of ESD or EMR according to risk stratification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESD (Active Comparator): Lesion with overt stigmata of SMIC or those with high risk (=> 10%) for covert SMIC.
  Interventions: Procedure: Endoscopic Submucosal Dissection
- EMR (Active Comparator): Lesion with no overt or a low risk for (<10%) for covert SMIC
  Interventions: Procedure: Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection — Endoscopic Submucosal Dissection (ESD) results in en-bloc resection of LSL, regardless of lesion size. This allows for accurate histopathological assessment of SMIC, R0/R1 resection and depth of invasion. ESD is considered a potentially curative for superficial cancers (T1a).
  Other Names: ESD
  Arms: ESD
Procedure: Endoscopic Mucosal Resection — EMR is the current standard for treating colonic LSL and has been validated to be safe and efficacious. LSLs => 20mm are frequently resected piecemeal. Recent research show that resection margin soft coagulation reduces recurrence rates to those similar to en-bloc resections.
  Other Names: EMR
  Arms: EMR

SUMMARY:
Colonic Laterally spreading lesions (LSL) => 20mm are at high risk to progress to cancer. Overt stigmata of submucosal invasive cancer (SMIC) has been well characterized and includes ulceration and surface pit pattern changes as per the Kudo classification of type V.

In a recent report, risk factors for LSL with SMIC and no overt stigmata (i.e. covert SMIC) were described. Resection of these lesions 'en-bloc' can allow for better histological staging and potentially reduce the need for surgical resection.

DETAILED DESCRIPTION:
With over 14,000 patients diagnosed annually, colorectal carcinoma (CRC) is the second most frequently invasive malignancy in Australia. By not only diagnosing CRC at an early stage, but also removing precursor adenomas, colonoscopy with polypectomy reduces the risk of developing and dying from CRC.

Laterally spreading lesions >= 20mm (LSL) are more likely to progress to cancer. The prevalence of LSL ranges from 1-5% in screening population. The risk of malignant progression of colorectal adenomas found during colonoscopy increases with lesion size, i.e. the cancer preventive effect is likely to be maximal in large lesions. Patients with LSL have a higher risk of malignancy and a higher recurrence rate of adenoma after lesion removal compared with diminutive polyps.

Endoscopic imaging can now accurately predict LSL with submucosal invasive cancer (SMIC) through assessment of LSLs morphology (Paris classification, granularity) and surface pit-pattern (Kudo classification). Such cases can be considered to have LSL with overt risk of SMIC.

Recent publication has highlighted that some LSLs might hrbor SMIC without overt morphological features (i.e. high risk for covert SMIC). These LSL with high risk of covert SMIC stratified LSLs based on lesion location and lesion morphology.

Generally LSLs can be safely and effectively removed by wide field endoscopic mucosal resection (WF-EMR) in over 90% of cases in competent hands.

One of the draw backs with WF-EMR is it requires piecemeal resection and thus is limited in providing assessment of complete excision and depth of submucosal invasion in cases where SMIC is present.

Thus, endoscopic en-bloc resection is preferable from an oncologic standpoint to obtain a single specimen for proper histopathologic assessment. Endoscopic submucosal dissection (ESD) is a technique that is now becoming the preferred method for achieving a complete endoscopic and histologic resection, referred to as R0. Evidence from retrospective cohort and meta-analyses suggests ESD provides a more consistent oncologic resection with a reduced rate of recurrence. However, the major limitations with the technique relate to increased procedure time and the skill-set required for performing the procedure.

One of the other major limitations of ESD is significant cost associated with the procedure, which includes procedure time and additional equipment in addition to the treatment of any subsequent complications. As such the implementation of ESD as the standard of care for all colorectal lesions has not been undertaken in Western countries, however it may have an important role for selective cases especially where there is concern for sub-mucosal invasive cancer (SMIC).

The investigators propose a selective ESD strategy to be performed for patients focusing on overt evidence of SMIC and those at high risk of covert SMIC (defined as risk >10%). The investigators will follow a prospective cohort study assessing the use of selective ESD strategy in the colorectum in the Western population.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for colorectal resection of large laterally spreading lesions in colon.
* Can give informed consent to trial participation

Exclusion Criteria:

* Previous resection or attempted resection of target adenoma lesion
* Endoscopic appearance of invasive malignancy
* Age less than 18 years
* Pregnancy
* Active Inflammatory colonic conditions (e.g. inflammatory bowel disease)
* Use of anticoagulant or antiplatelet agents other than aspirin outside of internationally recognised guidelines
* American Society of Anesthesiology (ASA) Grade IV-V

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Estimated)
Dates: Start 2017-08-14 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Rate of surgical referral | 3 months post procedure
  Incidence of surgical referral due to non-curative endoscopic resection.

SECONDARY OUTCOMES:
R0 resection rate | 3 months post procedure
  Rate of en-bloc resection with clear resection margins.
En Bloc resection rate | 3 months post procedure
  Rate of en-bloc resection
Technical success rate | 3 months post procedure
  Rate of procedures completed as per protocol
Duration of procedure | procedure
  Procedure duration in minutes.
Adenoma recurrence rate | 3 years post procedure
  Rate of recurrent adenoma at resection site on follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Result] Zauber AG, Winawer SJ, O'Brien MJ, Lansdorp-Vogelaar I, van Ballegooijen M, Hankey BF, Shi W, Bond JH, Schapiro M, Panish JF, Stewart ET, Waye JD. Colonoscopic polypectomy and long-term prevention of colorectal-cancer deaths. N Engl J Med. 2012 Feb 23;366(8):687-96. doi: 10.1056/NEJMoa1100370. PMID 22356322
- [Result] Iishi H, Tatsuta M, Iseki K, Narahara H, Uedo N, Sakai N, Ishikawa H, Otani T, Ishiguro S. Endoscopic piecemeal resection with submucosal saline injection of large sessile colorectal polyps. Gastrointest Endosc. 2000 Jun;51(6):697-700. doi: 10.1067/mge.2000.104652. PMID 10840302
- [Result] Risio M. The natural history of colorectal adenomas and early cancer. Pathologe. 2012 Nov;33 Suppl 2:206-10. doi: 10.1007/s00292-012-1640-6. PMID 22945585
- [Result] Moss A, Bourke MJ, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Chen RY, Byth K. Endoscopic mucosal resection outcomes and prediction of submucosal cancer from advanced colonic mucosal neoplasia. Gastroenterology. 2011 Jun;140(7):1909-18. doi: 10.1053/j.gastro.2011.02.062. Epub 2011 Mar 8. PMID 21392504
- [Result] Nanda KS, Tutticci N, Burgess NG, Sonson R, Williams SJ, Bourke MJ. Endoscopic mucosal resection of laterally spreading lesions involving the ileocecal valve: technique, risk factors for failure, and outcomes. Endoscopy. 2015 Aug;47(8):710-8. doi: 10.1055/s-0034-1391732. Epub 2015 Mar 12. PMID 25763831
- [Result] Oka S, Tanaka S, Saito Y, Iishi H, Kudo SE, Ikematsu H, Igarashi M, Saitoh Y, Inoue Y, Kobayashi K, Hisabe T, Tsuruta O, Sano Y, Yamano H, Shimizu S, Yahagi N, Watanabe T, Nakamura H, Fujii T, Ishikawa H, Sugihara K; Colorectal Endoscopic Resection Standardization Implementation Working Group of the Japanese Society for Cancer of the Colon and Rectum, Tokyo, Japan. Local recurrence after endoscopic resection for large colorectal neoplasia: a multicenter prospective study in Japan. Am J Gastroenterol. 2015 May;110(5):697-707. doi: 10.1038/ajg.2015.96. Epub 2015 Apr 7. PMID 25848926
- [Result] Lee EJ, Lee JB, Lee SH, Youk EG. Endoscopic treatment of large colorectal tumors: comparison of endoscopic mucosal resection, endoscopic mucosal resection-precutting, and endoscopic submucosal dissection. Surg Endosc. 2012 Aug;26(8):2220-30. doi: 10.1007/s00464-012-2164-0. Epub 2012 Jan 26. PMID 22278105
- [Result] Terasaki M, Tanaka S, Oka S, Nakadoi K, Takata S, Kanao H, Yoshida S, Chayama K. Clinical outcomes of endoscopic submucosal dissection and endoscopic mucosal resection for laterally spreading tumors larger than 20 mm. J Gastroenterol Hepatol. 2012 Apr;27(4):734-40. doi: 10.1111/j.1440-1746.2011.06977.x. PMID 22098630
- [Result] Burgess NG, Hourigan LF, Zanati SA, Brown GJ, Singh R, Williams SJ, Raftopoulos SC, Ormonde D, Moss A, Byth K, Mahajan H, McLeod D, Bourke MJ. Risk Stratification for Covert Invasive Cancer Among Patients Referred for Colonic Endoscopic Mucosal Resection: A Large Multicenter Cohort. Gastroenterology. 2017 Sep;153(3):732-742.e1. doi: 10.1053/j.gastro.2017.05.047. Epub 2017 Jun 2. PMID 28583826